CLINICAL TRIAL: NCT02002754
Title: Randomised, Open-label, Parallel-group Study of the Response to Bronchodilator Treatment in Subjects With Eosinophilic Bronchitis and the Mechanism of Varied Responses to Bronchodilator Treatment.
Brief Title: The Effect of Bronchodilator on Eosinophilic Bronchitis and Cough Variant Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kefang Lai, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cough2009
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Eosinophilic Bronchitis; Cough Variant Asthma
Keywords: eosinophilic bronchitis; cough variant asthma; bronchodilator
MeSH Terms: conditions — Cough-Variant Asthma | interventions — bambuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eosinophilic bronchitis (Active Comparator): Bambuterol Hydrochloride tablets 10mg,QN,for 3 days
  Interventions: Drug: Bambuterol Hydrochloride tablets
- cough variant asthma (Active Comparator): Bambuterol Hydrochloride tablets 10mg,QN,for 3 days
  Interventions: Drug: Bambuterol Hydrochloride tablets

INTERVENTIONS:
Drug: Bambuterol Hydrochloride tablets — Bambuterol Hydrochloride tablets(10mg) 3 tablets qd for three days(swallowed by warm water at 0.5-1h after each meal)

SUMMARY:
This study aim is to observe the response to Bambuterol Hydrochloride tablets treatment in subjects with eosinophilic bronchitis .

The investigators hypothesize:

A few of subjects with EB have some responses to Bambuterol Hydrochloride tablets therapy.

Most of subjects with CVA respond well to Bambuterol Hydrochloride tablets therapy

DETAILED DESCRIPTION:
Study groups:

45 patients with chronic cough will be collected and two groups will formed based on diagnosis as follows:

Group 1: EB group The patients with eosinophilic bronchitis received Bambuterol Hydrochloride tablets 10mg Q24 for three days .

Group 2: CVA group The patients with cough variant asthma received Bambuterol Hydrochloride tablets 10mg Q24 for three days .

Observe the response to Bambuterol Hydrochloride tablets treatment three days later and compare the effective rate of patients with EB and CVA. Then the study will be over.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a history of cough as sole or main symptom lasting more than 8 weeks.
2. Patients whose chest x-ray outcome was normal or without any active focus.
3. Patients with eosinophilic bronchitis who were diagnosed with the result of sputum eosinophil percentage (Eos%) over 2.5%, and the negative result in bronchial provocation test by methacholine inhalation challenge.
4. Patients with cough variant asthma have positive result in bronchial provocation test.
5. Patients who was aged from 18 years old (≥ 18 years old ) to 75 years old (≤ 75 years old).

Exclusion Criteria:

1. Patients who is a smoker or ex-smoker and has smoked within the previous year or has a cumulative smoking history >10 pack-years or equivalence.
2. Patients with concomitance of GERC (gastroesophageal reflux-related chronic cough), chronic bronchitis , bronchiectasis, bronchial tuberculosis, ACEI induced cough, bronchogenic carcinoma, psychologic cough, pulmonary fibrosis, bronchus foreign body, microlithiasis, tracheobroncheopathia osteochondroplastica, mediastinal tumor, left ventricular dysfunction.
3. Female subjects who are pregnant, breast-feeding or risk of becoming pregnant during the study.
4. Subjects who are diagnosed with past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease. e.g.nasal-sinus infection, lower respiratory tract infection, chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis or bronchopulmonary dysplasia.
5. Subjects who demonstrate significant abnormality on biochemistry, hematology, ECG.
6. Patients who does not cooperate with us.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Day-time and night-time cough symptom total-score changes from baseline to day 3. | three days

SECONDARY OUTCOMES:
cough sensitivity from baseline to day 3 | three days

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China